CLINICAL TRIAL: NCT05572047
Title: Coherent Sine Burst (CSE) Electroporation System Pilot Study in Patients With Atrial Fibrillation
Acronym: BURST-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arga Medtech SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP CSR 01-2022
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ablation; Coherent Sine-Burst; Electroporation; CSE
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Non-randomized, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Coherent Sine-Burst Electroporation for AF (Experimental): Patients with paroxysmal AF will receive treatment using the Arga Medtech Coherent Sine-Burst Electroporation ablation system to achieve pulmonary vein isolation (plus cavo-tricuspid isthmus ablation as necessary)
  Patients with persistent AF will receive treatment using the Arga Medtech Coherent Sine-Burst Electroporation ablation system to achieve pulmonary vein isolation and posterior wall ablation (and cavo-tricuspid isthmus ablation as necessary)
  Interventions: Device: Arga Medtech Coherent Sine-Burst Electroporation (CSE) Ablation System

INTERVENTIONS:
Device: Arga Medtech Coherent Sine-Burst Electroporation (CSE) Ablation System — Use of coherent sine-burst electroporation to ablate paroxysmal and persistent AF
  Other Names: CSE

SUMMARY:
To evaluate the safety and efficiency of the Arga Medtech CSE Ablation System in the treatment of atrial fibrillation.

DETAILED DESCRIPTION:
A prospective, single-arm, multi-center, multi-national, non-randomized study designed to provide clinical data to support the use of the Arga Medtech System in the ablation of atrial fibrillation.

Patients with paroxysmal AF will be treated using the Arga Medtech System to achieve pulmonary vein isolation (PVI) (and cavo-tricuspid isthmus (CTI) ablation as appropriate if history of CTI flutter or inducible flutter during procedure)

Patients with persistent AF will be treated using the Arga Medtech System to achieve PVI and posterior wall (PW) ablation (CTI ablation as above).

Patients will be remapped at 90 days post the index procedure to confirm absence of PV reconnection and durability of any additional lesion sets performed. Re-ablation is permitted during the remapping procedure if indicated. Re-ablation resets the 90-day blanking period.

Additional follow-ups will be conducted at 7 days, 30 days, 180 days and 360 days post the index or re-ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for ablation of paroxysmal or persistent AF
* Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the duration of the study
* Willing and able to give informed consent
* Failed at least one antiarrhythmic drug (AAD) (Class I to IV) as evidenced by recurrent symptomatic AF or intolerable or contraindicated to the AAD

Exclusion Criteria:

* Contraindication to AF ablation, TEE or anticoagulation
* Duration of continuous AF lasting longer than 12 months
* History of previous LA ablation or surgical treatment of AF/AT/AFL
* AF secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause
* Structural heart disease described as:

  * LVEF <30% based on TTE within 6 months of procedure
  * Left atrial size > 50mm based on TTE within 6 months of procedure (parasternal view)
* An implanted pacemaker or ICD
* Previous cardiac surgery, ventriculotomy, or atriotomy (excluding atriotomy for CABG)
* Previous cardiac valvular surgical or percutaneous procedure or prosthetic valve
* Interatrial baffle, closure device, patch, ASD or PFO
* Presence of a left atrial appendage occlusion device
* CABG or PTCA procedure within the last 6 months
* Unstable angina or ongoing myocardial ischemia
* Myocardial infarction within the previous 6 months
* Hypertrophic cardiomyopathy defined as left ventricular septal wall thickness > 1.5cm
* History of blood clotting or bleeding disease
* Prior history within the previous 6 months of documented cerebral infarction, TIA or system embolism
* Pregnant or lactating (current or anticipated within study follow-up)
* Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcomes measurement for this study
* Any other condition, in the judgment of the investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Serious system and procedure-related events | Within one week (7 days) post-procedure)
  Incidence of system-related and procedure-related serious adverse events (SAEs).
Procedural Success | Acute and/or up to 90 days post procedure
  Number of patients that achieve procedural success defined as isolation of the pulmonary veins at the index or re-mapping procedure.
Chronic isolation of the pulmonary veins | 90 to 180 days post index procedure
  Rate of patients and targeted pulmonary veins with documented electrical isolation of the pulmonary veins, assessed by entrance and exit block during a mapping procedure ~90-days post procedure.

SECONDARY OUTCOMES:
Freedom from documented atrial fibrillation (AF) | Up to 455 days post-index procedure
  Proportion of patients free from documented AF > or = 30 seconds of AF during follow-up.
Freedom from documented atrial arrhythmias (AF, AT and AFL) | Up to 455 days post-index procedure
  Freedom from documented atrial arrhythmias (AF, AT and AFL) > or = to 30 seconds during follow-up.
Freedom from documented symptomatic recurrence of atrial arrhythmias | Up to 455 days post-index procedure
  Freedom from recurrence of documented atrial arrhythmias (AF, AT and AFL) > or = to 30 seconds during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ante Anic, MD, Principal Investigator — University Hospital of Split; Giorgi Papiashvili, Principal Investigator — Israeli-Georgian Medical Research Clinic Helsicore
Locations (3):
- Croatia (2):
  - University Hospital of Split, Split
  - KBC Zagreb, Zagreb
- Israeli-Georgian Medical Research Clinic Helthycore Ltd, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anic A, Velagic V, Papiashvili G, Sikiric I, Lorenzo M, Prepolec I, Aranza I, Kapanadze N, Dagelic M, Breskovic T, Jurisic Z. Sine wave electroporation in patients with atrial fibrillation: Initial results of the BURST-AF study. Heart Rhythm. 2025 Aug;22(8):1946-1956. doi: 10.1016/j.hrthm.2025.04.042. Epub 2025 Apr 26. PMID 40294734